CLINICAL TRIAL: NCT06929520
Title: The Development and Evaluation of a Culturally Grounded ENDS Intervention for Rural Hawaiian Youth
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: University of California, Riverside (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: R01DA054215 (NIH)
Record Dates: First submitted 2025-04-07; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: E-cigarette Use; Substance Use
MeSH Terms: conditions — Vaping; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Dynamic wait-listed control group design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ENDS Prevention Intervention (Experimental): Participants will receive the ENDS Prevention Intervention consisting of (1) a modular classroom curriculum, (2) social media content, and (3) print media campaign.
  Interventions: Behavioral: ENDS Prevention Intervention (TBD)
- Treatment-as-usual control (No Intervention): Participants will receive treatment-as-usual, which consists of the standard health curriculum delivered in public schools.

INTERVENTIONS:
Behavioral: ENDS Prevention Intervention (TBD) — The ENDS Prevention Intervention will consist of (1) a modular classroom curriculum with ENDS-focused lessons and lessons covering alcohol, tobacco, and other drug use; (2) social media content that is related to the classroom curriculum and video content, and (3) a print media campaign across school campuses on Hawaii Island.
  Arms: ENDS Prevention Intervention

SUMMARY:
The purpose of this research proposal is to develop and evaluate a culturally grounded, ENDS prevention intervention for rural Hawaiian youth. This will be accomplished through two specific aims. AIM 1 (Years 1-3) are focused on pre-intervention and intervention development. In Year 1, youth focus groups will be conducted to assess the environmental demands related to ENDS use in rural Hawai'i. In Year 2, specific ENDS-related problem situations (i.e., situations that increase risk for ENDS use) will be extracted from the Year 1 focus groups and prioritized through survey methods with 200-250 predominately Native Hawaiian youth across 16 different middle/intermediate schools on Hawai'i Island. In Year 3, five situations found to be the most frequently experienced and/or difficult to manage by youth surveyed in Year 2 will serve as the foundation for the development of narrative scripts. Three of these scripts will be cast and filmed on location on Hawai'i Island by a professional film director, and will be edited into three short films, 6-8 video clips, and 6-8 professional photos or production stills. Similar to the investigators' prior drug prevention research in rural Hawai'i, classroom-based lessons will be created to support the short films. Additional lessons and videos from an evidence-based, culturally grounded substance abuse prevention curriculum for Hawaiian youth (Ho'ouna Pono) will be used to create a modular classroom curriculum. The video clips and professional photography/production stills will be embedded with prevention messaging, and will be used for a social and print media campaign to reinforce the classroom curriculum. AIM 2 (Years 4-5) is to evaluate the ENDS prevention intervention (classroom curriculum plus social/print media campaign) across all middle/intermediate public or public-charter schools (N = 16) and up to 11 different cultural immersion charter schools on Hawai'i Island using a dynamic wait-listed control group design.

DETAILED DESCRIPTION:
Assessing Environmental Demands (Year 1). A qualitative design using focus groups and follow-up in-depth interviews will be used to examine the social, cultural, and developmental context of youth ENDS and dual use in rural Hawai'i. Ten to fifteen youth focus groups (3-5 members per group) will be conducted to identify problematic social situations involving offers to use ENDS (with or without combustible cigarettes) from peers, cousins, and adult family members. Participants will be asked to describe social situations where they encountered ENDS (with or without combustible cigarettes) being offered to them or where there was an implicit demand to use these substances. A convenience sample of Native Hawaiian youth participants will be recruited from at least sixteen rural public middle, intermediate, or multi-level schools on Hawai'i Island. Focus groups will be gender-specific, and group facilitators will match the gender of the groups.

Situation Identification and Prioritization (Year 2). The goal of this step is to operationalize and prioritize problematic social situations involving ENDS and dual use, by assessing them for their frequency of exposure and perceived difficulty for refusal. Fifty to one-hundred twenty-five potential items will be drawn from the focus group and interview data in Year 1, which will be reduced in number through expert analysis, and then be subjected to an assessment of social validity. The latter step entails youth participants rating each item on two criteria using Likert scales: (1) the frequency with which the subject encountered the situation (from never to more than 4 times per month), and (2) the perceived difficulty in dealing with the situation (from very easy to very difficult). The survey will be administered to 200-250 predominantly Native Hawaiian and Pacific Islander adolescents on Hawai'i Island. Descriptive statistics will be used to examine the prevalence of situations and their perceived difficulty. Exploratory factor analytic procedures will be used to establish subscales, and construct validity will be assessed by examining the relationship of the items to the use of ENDS and combustible cigarettes. Five of the most frequently experienced and/or challenging situations identified by surveyed youth will be translated into narrative scripts by a professional scriptwriter/videographer (Yamashita) in Year 3.

Video Production (Year 3). In this phase, five frequently experienced and difficult ENDS-related problem situations and youth-identified strategies to deal with them will be translated to a scripted format by an Emmy award-winning scriptwriter/videographer (Matt Yamashita; see letter of support). These scripts will evolve from situations prioritized in Year 2, but based on the research literature, we anticipate that they will focus on the use of ENDS e-liquid flavors, marijuana vaping, and/or dual use (ENDS and combustible cigarette use). Three of the five scripts will be cast, filmed on location on Hawai'i Island, and edited into three 5-7 minute videos. Each will depict a main storyline, and three different endings demonstrating refusal strategies of varying levels of competence. This phase will not entail human subjects.

Lesson and Social/Print Media Development (Year 3). In this phase, three new ENDS prevention lessons will be developed that are focused on the videos, and will be delivered with 4 of 7 ATOD lessons developed and evaluated in the Ho'ouna Pono efficacy trial (R01 DA037836). These will be delivered as part of a modular prevention intervention, where teachers will be able to select the four Ho'ouna Pono lessons to accompany the three ENDS-focused lessons, in order to customize the curriculum to fit their students' needs. Social media components (i.e., short video clips with embedded ENDS prevention messaging) and print media components (i.e., poster-sized still images with embedded ENDS prevention messaging) will also be created. The three ENDS prevention lessons and social/print media components will be validated by a sample of Native Hawaiian youth (n = 10-15) and educational stakeholders (n = 10-15). The classroom lessons will be delivered by teachers in participating schools as part of the health curriculum, while the social and print media components will be delivered concurrently with the classroom-based curriculum. The social media components will be delivered through popular social media platforms (Instagram, Snapchat, and/or TikTok) using school-supervised accounts, while the print media components will be posted on bulletin and message boards throughout schools receiving the intervention.

Efficacy Trial (Years 4-5). A dynamic wait-listed control group design will be employed to examine the longitudinal effects of the ENDS intervention (i.e., modular prevention curriculum and social/print media campaign). All participating schools will be block randomized based on region (north, south, east, and west Hawai'i) into four cohorts, and cohorts will be randomly assigned to receive the intervention at designated times staggered across the two-year evaluation period. Schools in Cohorts 1 and 2 will receive the intervention in Year 4 of the study, while schools in Cohorts 3 and 4 will receive the intervention in Year 5. As a result, all schools will be evaluated at pre-test and immediate post-test, and schools in Cohorts 1-3 will receive follow up evaluations. Schools in Cohort 1 will receive follow ups at 3-, 9-, 12-, and 15-months post-intervention, Cohort 2 at 6-, 9-, and 12-months post-intervention, and Cohort 3 at 3-months post-intervention. In terms of measurement, the survey used to evaluate the efficacy of the ENDS prevention intervention will include standard demographic items covering areas such as age, grade, gender, family structure, and SES, as well as 52 items related to culture/enculturation, risk and protective factors (including ENDS and combustible cigarette use frequency), resistance strategies, risk assessment, and peer affiliations. Main effects related to ENDS and dual use will be measured, as well as the use of different resistance strategies depicted in the videos. Peer affiliations over time will also be measured to examine the effect of the intervention on the social and relational context of youth in rural Hawai'i.

ELIGIBILITY:
Inclusion Criteria:

* 6th-8th grade students attending a public or public-charter school on Hawaii Island.

Exclusion Criteria:

* K-5th grade students and 9th-12th grade students on Hawaii Island.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2027-05-15 (Estimated); Study Completion 2027-05-15 (Estimated)

PRIMARY OUTCOMES:
Recent Electronic Nicotine Delivery System (ENDS) use | Up to 19 months
  Past 30-day use of e-cigarettes and/or vaping devices

SECONDARY OUTCOMES:
Recent Alcohol, Tobacco, and Other Drug (ATOD) use | Up to 19 months
  Past 30-day alcohol, tobacco, and other drug use

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hawaii, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data, consistent with the NIH Data Safety and Monitoring plan for this study, will be shared with other researchers upon request.